CLINICAL TRIAL: NCT00000679
Title: (Ro 24-2027) A Randomized, Double-Blind, Comparative Study of Dideoxycytidine (ddC) Versus Zidovudine (AZT) in Patients With AIDS or Advanced ARC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Hoffmann-La Roche (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 114; Protocol Number: N3300A; FDA 31A; Study Number: 3-27
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-03-14 (Estimated); Status verified 1994-12

CONDITIONS: HIV Infections
Keywords: Zalcitabine; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine; Zalcitabine

INTERVENTIONS:
Drug: Zidovudine
Drug: Zalcitabine

SUMMARY:
To show that zalcitabine (dideoxycytidine; ddC) is at least as effective as zidovudine (AZT) in the treatment of AIDS or advanced AIDS related complex (ARC), and also that ddC shows a different safety profile than AZT.

In clinical studies, ddC shows antiviral activity. Because of the antiviral activity, and because of the low incidence of mild, reversible neurotoxicity and absence of blood-related toxicity with low dose ddC therapy, a long-term Phase II/III study comparing ddC to AZT in patients with AIDS or advanced ARC is now warranted.

DETAILED DESCRIPTION:
In clinical studies, ddC shows antiviral activity. Because of the antiviral activity, and because of the low incidence of mild, reversible neurotoxicity and absence of blood-related toxicity with low dose ddC therapy, a long-term Phase II/III study comparing ddC to AZT in patients with AIDS or advanced ARC is now warranted.

After screening, physical examination and laboratory tests (within 14 days of entry) patients are randomized to one of two treatment groups. They receive either ddC plus an AZT placebo or AZT plus a ddC placebo. Because it is a blinded study, patients do not know which group they are in. Patients are evaluated weekly for the first 10 weeks and then biweekly thereafter.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Aerosolized pentamidine (300 mg once every 4 weeks) for Pneumocystis carinii pneumonia (PCP) prophylaxis.
* Neuroleptics, benzodiazepines, or antidepressants if patient has been stable with chronic treatment > 1 month.
* Low dose benzodiazepines or low dose antidepressants.
* Drugs that are unlikely to cause increased toxicity with either study drug and are unlikely to cause peripheral neuropathy.
* Drugs with little nephrotoxicity, hepatotoxicity, or cytotoxicity that the patient has been taking and tolerating well.
* Acyclovir (up to 600 mg/kg/day) for up to 21 days.
* Ketoconazole (up to 400 mg/day) Nystatin.
* Low-dose acetaminophen or nonsteroidal anti-inflammatory agents.
* Isoniazid if patient has no evidence of peripheral neuropathy at entry and if patient takes 50 mg/day pyridoxine concomitantly with isoniazid.
* Allowed with interruption of study medication for up to 21 days per episode and for a total of 42 days for the study:
* Drugs that could cause serious additive toxicity when coadministered with either study medication for treatment of an acute intercurrent illness or opportunistic infection, including:
* Acyclovir (< 600 mg/day), fluconazole, systemic pentamidine, foscarnet, pyrimethamine, triple sulfa, ansamycin, ganciclovir, trimethoprim / sulfamethoxazole.

Patients must have a diagnosis of AIDS or advanced AIDS related complex (ARC). At least 20 percent of the patients must have a consistently positive serum HIV p24 antigen (= or > 70 pg/ml) as defined by the Abbott HIV antigen test, on two separate occasions at least 72 hours apart.

* Patients found at screening to have a temperature > 38.5 degrees C should be evaluated for the possibility of an occult opportunistic or bacterial infection or neoplasm. If this complete evaluation reveals an infection, they can be entered. If this evaluation is unrevealing, they may be entered after evaluation is completed but while mycobacterial cultures are still pending. Patients with a history of unexplained temperatures > 38.5 degrees C should be evaluated as above and/or be afebrile (temperature < 38.0 degrees C) for 2 weeks prior to study entry.
* Allowed: Kaposi's sarcoma not specifically excluded, basal cell carcinoma of the skin or in situ carcinoma of the cervix.
* Current positive venereal disease research label (VDRL) and fluorescent treponemal antibody (FTA) if treated as for asymptomatic neurosyphilis.

Prior Medication:

Allowed:

* Drugs that cause peripheral neuropathy and drugs that could cause significant increased toxicity with zidovudine (AZT) or dideoxycytidine (ddC) including experimental drugs if therapy with these drugs is completed and patient is stable for 14 days.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Active AIDS defining opportunistic infection or other active intercurrent illness is excluded if ongoing treatment requires the use of excluded concomitant medication.
* Patients with symptomatic visceral Kaposi's sarcoma (KS), progression of KS within the month prior to entry into the study, or with current neoplasms not specifically allowed.
* Severe AIDS dementia complex defined by a score of < 23 on the Mini-Mental State Exam.
* Signs, symptoms, or history of peripheral neuropathy.
* Significant cardiac disease, defined as history of ventricular arrhythmias requiring medication, prior myocardial infarct, or history of angina or ischemia changes on ECG (electrocardiography).
* Requiring > 2 weeks of acyclovir therapy at > 600 mg/day.
* Current positive venereal disease research label (VDRL) and fluorescent treponemal antibody (FTA) not specifically allowed.
* Significant liver disease.

Concurrent Medication:

Excluded:

* Drugs that cause peripheral neuropathy:
* chloramphenicol, cisplatinum, iodoquinol, dapsone, phenytoin, disulfiram, ethionamide, glutethimide, gold, hydralazine, ribavirin, metronidazole, vincristine, nitrofurantoin.
* Drugs that could cause significant increased toxicity with zidovudine (AZT) or dideoxycytidine (ddC), including experimental drugs not specifically allowed.
* Drugs that could cause seizures or changes in mental status or neurological examination.

Concurrent Treatment:

Excluded:

* Transfusion dependency.

Patients with the following are excluded:

* Active AIDS defining opportunistic infection or other active intercurrent illness if ongoing treatment requires use of excluded concomitant medication.
* Symptomatic visceral Kaposi's sarcoma (KS), progression of KS within the month prior to study entry, or current neoplasms not specifically allowed.
* Severe AIDS dementia complex defined by a score of < 23 on the Mini-Mental State Exam.
* Signs, symptoms, or history of peripheral neuropathy.
* Unwilling or unable to sign informed consent.

Prior Medication:

Excluded:

* Zidovudine (AZT), dideoxycytidine (ddC), or any other antiretroviral nucleoside analog.
* Excluded within 90 days of study entry:
* Any experimental drug including fluconazole, ganciclovir, foscarnet, erythropoietin, or ribavirin.

Excluded within 90 days of study entry:

* Drugs that have caused significant nephrotoxicity or significant hepatotoxicity.
* Drugs that could cause peripheral neuropathy including phenytoin, hydralazine, metronidazole, and nitrofurantoin.
* Systemic corticosteroids or immunomodulators including interferon and interleukin.

Prior Treatment:

Excluded within 30 days of study entry:

* Radiation therapy.

Active substance or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Primary Completion 1994-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Kaiser Foundation Hosp, Harbor City, California
  - Kaiser Permanente Med Ctr, Los Angeles, California
  - UCD Med Ctr, Sacramento, California
  - Davies Med Ctr, San Francisco, California
  - Mount Zion Med Ctr, San Francisco, California
  - San Francisco Veterans Administration Med Ctr, San Francisco, California
  - Santa Clara Valley Med Ctr, San Jose, California
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Ctr for Special Immunology, Fort Lauderdale, Florida
  - Comprehensive Clinic / Dr Robert Schwartz, Fort Myers, Florida
  - Med Service, Miami, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Northwestern Univ Med School, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - New England Med Ctr, Boston, Massachusetts
  - Henry Ford Hosp, Detroit, Michigan
  - Saint Michael's Med Ctr, Newark, New Jersey
  - Albany Med College / AIDS Treatment Ctr, Albany, New York
  - Sunset Park Health Ctr - Lutheran Med Ctr, Brooklyn, New York
  - Bowman Gray School of Medicine / North Carolina Baptist Hosp, Winston-Salem, North Carolina
  - Univ Hosp of Cleveland / Case Western Reserve Univ, Cleveland, Ohio
  - Graduate Hosp, Philadelphia, Pennsylvania
  - N Texas Ctr for AIDS & Clin Rsch, Dallas, Texas
  - Univ TX Galveston Med Branch, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Background] Bozzette SA, Hays RD, Berry SH, Kanouse DE. A Perceived Health Index for use in persons with advanced HIV disease: derivation, reliability, and validity. Med Care. 1994 Jul;32(7):716-31. doi: 10.1097/00005650-199407000-00005. PMID 8028406
- [Background] Bozzette SA, Hays RD, Berry SH, Kanouse DE, Wu AW. Derivation and properties of a brief health status assessment instrument for use in HIV disease. J Acquir Immune Defic Syndr Hum Retrovirol. 1995 Mar 1;8(3):253-65. doi: 10.1097/00042560-199503010-00006. PMID 7859137
- [Background] Bozzette SA, Kanouse DE, Berry S, Duan N. Health status and function with zidovudine or zalcitabine as initial therapy for AIDS. A randomized controlled trial. Roche 3300/ACTG 114 Study Group. JAMA. 1995 Jan 25;273(4):295-301. PMID 7815656
- [Background] Bozzette SA, Kanouse D, Berry S, Duan N, Downes-LeGuin T, Hays R, Petinnelli C, Richman DD, Gocke D, Kahn J. Relative effects of ddC or ddI versus ZDV on health status, function and disability in N3300 (ACTG 114) and ACTG 116b/117. Int Conf AIDS. 1992 Jul 19-24;8(1):Mo21 (abstract no MoB 0077)
- [Background] Remick S, Follansbee S, Olson R, Pollard R, Reiter W, Salgo M. Safety and tolerance of zalcitabine (ddC, HIVID) in a double-blind, comparative trial (ACTG 114; N3300). Int Conf AIDS. 1993 Jun 6-11;9(1):488 (abstract no PO-B26-2115)
- [Background] Follansbee S, Drew L, Olson R, Pollard R, Relter W, Salgo M. The efficacy of zalcitabine (ddC, HIVID) versus zidovudine (ZDV) as monotherapy in ZDV naive patients with advanced HIV disease: a randomized, double-blind, comparative trial (ACTG 114; N3300). Int Conf AIDS. 1993 Jun 6-11;9(1):487 (abstract no PO-B26-2113)
- [Background] Gries JM, Troconiz IF, Verotta D, Jacobson M, Sheiner LB. A pooled analysis of CD4 response to zidovudine and zalcitabine treatment in patients with AIDS and AIDS-related complex. Clin Pharmacol Ther. 1997 Jan;61(1):70-82. doi: 10.1016/S0009-9236(97)90183-1. PMID 9024175